CLINICAL TRIAL: NCT01610648
Title: Improving the Sensitivity and Specificity of the STOP-Bang Screening Questionnaire for Patients With Obstructive Sleep Apnea
Brief Title: Improving the STOP-Bang Screening Questionnaire for Patients With Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IRB#10391
Record Dates: First submitted 2012-05-23; First posted 2012-06-04 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Sleep Apnea; Metabolic Syndrome
Keywords: OSA; metabolic syndrome; Apnea-hypopnea index; Oxygen desaturation index
MeSH Terms: conditions — Sleep Apnea Syndromes; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients presenting for a diagnostic sleep study: Patients presenting to the TMC sleep center for sleep study

SUMMARY:
The study is being conducted to test the ability of a simple questionnaire to detect mild, moderate or severe obstructive sleep apnea. The investigators are also investigating whether adding the size of the neck and waist can add to the accuracy of the questionnaire.

The study will be conducted at the Center for Sleep Medicine at Tufts Medical Center. The investigators hope to enroll 250 patients in our study at Tufts Medical Center.

DETAILED DESCRIPTION:
We will complete a 12 item questionnaire and data sheet with the study subjects based on their responses and 2 measurements specified below, right before application of a study the start of their sleep study called "Polysomnography".

If available, we will also use information from the subjects medical record, including information regarding a history of diabetes (blood sugar that is too high), high blood pressure and laboratory data such as blood sugar and blood lipids (fats in the blood). We will record this information for research purposes.

The 2 measurements performed for research purposes consist of the size of the neck and waist using a flexible tape measure. After the sleep study, we will also use results from that study in this research. We expect the subjects study participation to be completed in 30 minutes or less.

There will be no follow up. If a participant cannot complete the sleep study for any reason, the study team may decide to withdraw the subject's participation without further notice.

The study will be open for participation from June 2012 through November of 2012.

ELIGIBILITY:
Inclusion Criteria:

* Referral to the sleep center for a diagnostic study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting for a sleep study to Tufts Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Cut-off value determination for each of three STOP-Bang versions | The outcome measure will be assessed after aggregate data analysis has been completed. It is expected for January 2013 (up to 2 years)
  Determine the best cutoff value using receiver-operating characteristics curves separately for each of the 3 versions of the STOP-Bang questionnaire (original, re-weighted, Stop-Bang MEtS) for subjects with confirmed mild, moderate and severe sleep apnea according to the Apnea-Hypopnea Index AHI as defined by the society for sleep medicine. The cut-off values will be calculated separately for each category of severity.

SECONDARY OUTCOMES:
Cut-off value determination for each of three STOP-Bang versions | The outcome measure will be assessed after aggregate data analysis has been completed. It is expected for January 2013 (up to 2 years)
  Determine the best cutoff value using receiver-operating characteristics curves separately for each of the 3 versions of the STOP-Bang questionnaire (original, re-weighted, Stop-Bang MEtS) for subjects with confirmed mild, moderate and severe sleep apnea according to the Oxygen Desaturation Index ODI as defined by the Society for sleep medicine. The cut-off values will be calculated separately for each category of severity.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Schumann, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Sleep Center, Tufts Medical Center, Boston, Massachusetts, United States